CLINICAL TRIAL: NCT05530031
Title: UBM Guided Site and Extent of Trabeculotomy in Pediatric Glaucoma
Acronym: UBM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Dina abdelfattah, Dina Abd Elfattah, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R.22.09.1801
Record Dates: First submitted 2022-09-03; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Glaucoma Pediatric
MeSH Terms: interventions — Trabeculectomy

STUDY DESIGN:
Intervention Model Description: • trabeculotomy (with Metal Trabeculotome): a scleral flap is raised at the selected site with UBM and a cutdown in shlemm's canal is performed, a metal trabeculotome is used to cannulate and tear through a section of the inner wall of SC and trabeculum into the AC. Closure of the scleral flap and conjunctiva with 10/0 nylon. Viscoelastic is used to dilate the schlemm's canal, form the anterior chamber and decrease the risk of hyphema.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pediatric glaucoma patients either primary or secondary (Experimental): All Cases with pediatric glaucoma prepared for trabeculotomy including Primary congenital glaucoma and secondary glaucoma as : glaucoma following cataract surgery and traumatic glaucoma
  Interventions: Procedure: trabeculotomy ( angle glaucoma surgery )

INTERVENTIONS:
Procedure: trabeculotomy ( angle glaucoma surgery ) — a scleral flap is raised at the selected site with UBM and a cutdown in shlemm's canal is performed, a metal trabeculotome is used to cannulate and tear through a section of the inner wall of SC and trabeculum into the AC. Closure of the scleral flap and conjunctiva with 10/0 nylon. Viscoelastic is used to dilate the schlemm's canal, form the anterior chamber and decrease the risk of hyphema.

SUMMARY:
Different types of surgery are applied in PCG, including goniotomy, trabeculotomy, glaucoma drainage devices and trabeculectomy. UBM examination of the anterior chamber before surgery can help in the decision to what type of surgery is best for the patient. Aim of the work To study the value of using UBM to select the site and extent of trabeculotomy in pediatric glaucoma and its correlation with surgical outcomes.

DETAILED DESCRIPTION:
To study the value of using UBM to select the site and extent of trabeculotomy in pediatric glaucoma and its correlation with surgical outcomes.All Cases with pediatric glaucoma prepared for trabeculotomy including Primary congenital glaucoma and secondary glaucoma as : glaucoma following cataract surgery and traumatic glaucoma Methods

History taking:

* Family history of ocular pathologies or syndromes.
* Age at which the mother noticed ocular affection, time and type of intervention.
* Onset of IOP elevation, IOP lowering medications used and any previous surgical intervention for glaucoma.

Preoperative examination & assessment

* Examination under anaesthesia for state of the conjunctiva, conreal incision scars, corneal diameter, Haab's stria, broad limbus, anterior chamber depth, regularity and content, pupil shape, centration and response to mydriatics, IOL position and status in pseudophakic cases, IOP value, optic nerve cupping.
* A scan for axial length and central corneal thickness.
* B scan ultrasonography.
* UBM : full detailed anterior segment examination will be done including : trabecular iris angle width , presence of abnormal iris insertion , abnormal membranes , Schlemm canal studying and iris thickness. All these parameters will be recorded for all 4 quadrants to select the most appropriate site of trabeculotomy.

Procedure

• trabeculotomy (with Metal Trabeculotome): a scleral flap is raised at the selected site with UBM and a cutdown in shlemm's canal is performed, a metal trabeculotome is used to cannulate and tear through a section of the inner wall of SC and trabeculum into the AC. Closure of the scleral flap and conjunctiva with 10/0 nylon. Viscoelastic is used to dilate the schlemm's canal, form the anterior chamber and decrease the risk of hyphema.

Follow up

* Postoperative visits planned on the first day, first week, second week, at first month, three months and six months.
* Outcome measures included the IOP value at each visit, corneal diameters, cup disc ratio if accessible, the number of glaucoma medications used, the number and kind of complications.
* Surgical success was defined as:

  1. Complete sucess when IOP >5mmHg and ≤21mmHg or 30% IOP reduction from baseline and without any further IOP-lowering surgery.
  2. Qualitative success when IOP ≤21mmHg or 30% IOP reduction from baseline but with the use of IOP lowering medications.
* Failure is defined as:
* IOP more than 21mmHg despite the use of IOP lowering medications.
* Hypotony: IOP ≤5mmHg persistent for more than two weeks.
* Need for other glaucoma surgery to control IOP.

ELIGIBILITY:
Inclusion Criteria:

- All Cases with pediatric glaucoma prepared for trabeculotomy including Primary congenital glaucoma and secondary glaucoma as : glaucoma following cataract surgery and traumatic glaucoma

Exclusion Criteria:

patients refusing the study

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure | 6 months
  success of glaucoma surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Dina Abd Elfattah, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
results